CLINICAL TRIAL: NCT06909149
Title: The Role of Amniotic Membrane Extract Eye Drops as an Adjunctive Therapy in Resistant Corneal Ulcers: A Randomized Clinical Trial Study
Brief Title: Role of Amniotic Membrane Extract Eye Drops as an Adjunctive Therapy in Resistant Corneal Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Sameh El-Shorbagy, Assistant Lecturer of Ophthalmology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33028/03/19
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Amniotic Membrane Extract Eye Drops; Resistant Corneal Ulcers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane extract eye drops group (Experimental): Patients received the amniotic membrane extract eye drops once every two hours during waking time as an adjunctive therapy to the specific treatment
  Interventions: Drug: Amniotic membrane extract eye drops
- Control group (Active Comparator): Patients received the specific treatment only
  Interventions: Drug: Specific treatment

INTERVENTIONS:
Drug: Amniotic membrane extract eye drops — Patients received the amniotic membrane extract eye drops once every two hours during waking time as an adjunctive therapy to the specific treatment.
  Arms: Amniotic membrane extract eye drops group
Drug: Specific treatment — Patients received the specific treatment only.
  Arms: Control group

SUMMARY:
This study aimed to assess the efficacy of amniotic membrane extract eye drops (AMEED) as a supplementary treatment for refractory corneal ulcers.

DETAILED DESCRIPTION:
Corneal ulceration is one of the leading causes of corneal blindness. Multiple causes of corneal ulceration vary in prevalence from country to country according to geographical and economic conditions.

Amniotic membrane (AM) contains pluripotent stem cells, highly organized collagen, immune-modulators, growth factors, anti-fibrotic and anti-inflammatory cytokines, A variety of matrix proteins, in addition to anti-microbial effect. Inspite of the amniotic membrane transplant is still a surgical procedure, it is not indicated in mild to moderate cases of resistant corneal ulceration and persistent epithelial defects and would alter visual function gravely.

Researchers found that amniotic membrane extract eye drops (AMEED) are superior to autologous blood serum in level and variety of growth factors, cytokines, and antimicrobial activity, along with higher success rates and faster healing results; they discarded the amniotic membrane conditioned medium as it failed to provide matching results.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 80 years.
* Both sexes.
* Patients who were suffering from corneal ulcers that showed no signs of improvement after one week of medical intervention.

Exclusion Criteria:

* Severe corneal melting.
* Perforated corneal ulcer.
* Corneal ulcers with significant thinning with or without descemetocele.
* Patients who were unable to adhere to the treatment plan properly.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Time of improvement of corneal ulcers | 7 weeks after the procedure
  Time of improvement of corneal ulcers will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.